CLINICAL TRIAL: NCT06283719
Title: A Phase I Dose Escalation Study of Tolerability, Safety, Efficacy, and Pharmacokinetics of ZG006 in Participants With Advanced Small Cell Lung Cancer or Neuroendocrine Carcinoma, Followed by a Phase II Dose Expansion Study in Participants With Advanced Small Cell Lung Cancer
Brief Title: Dose Escalation Study of ZG006 in Participants With Advanced Small Cell Lung Cancer or Neuroendocrine Carcinoma, Followed by Dose Expansion Study in Participants With Advanced Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZG006-002
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-12

CONDITIONS: Small Cell Lung Cancer; Neuroendocrine Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part1 ：Dose Escalation (Experimental): A total of six dose escalations were preset: 0.1 mg, 0.3 mg, 1 mg, 3 mg, 10 mg, and 30 mg.
  Interventions: Biological: ZG006
- Part2 ：Dose Expansion (Experimental): Part 2 consists of three cohorts. Cohort 1 is divided into two stages:
  Stage 1 is for dose optimization: approximately 30 patients will be enrolled in each of the two preliminary RP2D groups; the better-performing dose will be selected for Stage 2 based on emerging data.
  Stage 2 is the pivotal, registrational study, intended to enroll patients with advanced small-cell lung cancer who are in third-line or later lines of therapy.
  Interventions: Biological: ZG006

INTERVENTIONS:
Biological: ZG006 — ZG006 will be administered as an intravenous (IV) infusion.

SUMMARY:
This is a multicenter, open-label Phase I/II study consisting of two parts:

Part 1 is a Phase I dose-escalation study of ZG006, aimed at evaluating the safety and tolerability of ZG006 in Participants with advanced small-cell lung cancer or neuroendocrine carcinoma. Upon completion of Part 1, the investigators and sponsor will jointly determine two preliminary recommended Phase II doses for Part 2, based on the available safety, preliminary efficacy, and pharmacokinetic data.

Part 2 is a Phase II dose-expansion study of ZG006, designed to explore and confirm the efficacy and safety of ZG006 monotherapy in advanced small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form;
* Male or female 18~75 years of age;
* Eastern Cooperative Oncology Group(ECOG) Performance Status of 0 or 1;
* Life expectancy ≥ 3 months;
* Participants with histologically or cytologically confirmed advanced solid tumors who also fulfill the following: Part 1: advanced small-cell lung cancer (SCLC) or neuroendocrine carcinoma.Part 2: advanced SCLC.Specifically for Part 2 Cohort 1: de-novo SCLC (composite SCLC excluded).Stage 2 restricted to third-line or later.Cohort 2: transformed SCLC.Cohort 3: large-cell neuroendocrine carcinoma of the lung and composite SCLC.

Exclusion Criteria:

* Participants were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 2 years
  ORR is defined as the percentage of participants achieving a confirmed complete response (CR) or partial response(PR) based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 2 years
  The types and frequencies of adverse events (AEs) evaluated according to the National Cancer Institute Common Terminology Criteria for adverse events (NCI-CTCAE) version 5.0
Number of participants with serious adverse events (SAEs) | Up to approximately 2 years
Duration of response (DOR) | Up to approximately 2 years
  DOR is defined as the time from first evidence of response (CR or PR per RECIST 1.1) to earlier date of disease progression or death due to any cause
Disease control rate (DCR) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No